CLINICAL TRIAL: NCT00002792
Title: ALLOGENEIC MARROW OR PERIPHERAL BLOOD STEM CELL TRANSPLANTATION FOR AGNOGENIC MYELOID METAPLASIA WITH MYELOFIBROSIS
Brief Title: Combination Chemotherapy Plus Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Myeloproliferative Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1032.01; FHCRC-1032.01; NCI-H96-0929; CDR0000064859 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Myelodysplastic/Myeloproliferative Diseases
Keywords: polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Myelodysplastic-Myeloproliferative Diseases; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Busulfan; Cyclophosphamide; Cyclosporine; Methotrexate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining bone marrow or peripheral stem cell transplantation with chemotherapy may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus either bone marrow or peripheral stem cell transplantation in treating patients with myeloproliferative disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess disease free survival in patients with idiopathic myelofibrosis treated with a preparative busulfan/cyclophosphamide regimen followed by allogeneic bone marrow or peripheral blood stem cell transplantation.
* Determine the risk of primary graft failure in these patients.

OUTLINE: Patients receive a preparative regimen consisting of oral busulfan every 6 hours on days -7 through -4 and cyclophosphamide on days -3 and -2. Patients then receive allogeneic bone marrow or peripheral blood stem cells on day 0. Patients registered on protocol FHCRC-1106.00 randomized to stem cell transplant receive unmodified G-CSF-mobilized stem cells from an HLA-identical donor.

Patients receive cyclosporine/methotrexate or tacrolimus/methotrexate as prophylaxis for graft-versus-host disease (GVHD). Patients receiving marrow from unrelated donors are eligible for appropriate GVHD prophylaxis studies.

Patients are followed at 6 and 12 months after transplant.

PROJECTED ACCRUAL: A maximum of 20 patients will be accrued for this study over approximately 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Idiopathic myelofibrosis (IMF) with at least 1 poor prognosis characteristic, including but not limited to:

  * Hemoglobin less than 10 g/dL
  * Platelet count less than 100,000/mm^3
  * Hepatomegaly (i.e., palpable liver edge 5 cm below costal margin)
  * Clinical requirement for splenectomy
* Other myeloproliferative disorders in an IMF like myelofibrotic state eligible
* No evidence of leukemic progression, e.g.:

  * Greater than 15% peripheral blood blasts
  * Fever or bone pain of unknown origin
  * Rapidly progressing splenomegaly
* No other causes for myelofibrosis, such as:

  * Collagen vascular disorder
  * Lymphoma
  * Granulomatous infection
  * Metastatic carcinoma
  * Hairy cell leukemia
  * Myelodysplastic syndrome
* No active central nervous system disease
* One of the following donor/patient pairings is required:

  * Donor status:

    * Genotypic or phenotypic HLA-matched relative

      * Maximum patient age of 65
    * One antigen HLA-mismatched relative, HLA-matched unrelated donor, or one antigen HLA-mismatched unrelated donor

      * Maximum patient age of 55
* Transplant on this protocol allowed for patients registered on protocol FHCRC-1106.00

PATIENT CHARACTERISTICS:

Age:

* 65 and under

Performance status:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2 times normal
* SGPT no greater than 4 times normal

Renal:

* Creatinine no greater than two times normal OR
* Creatinine clearance at least 50%

Cardiovascular:

* Ejection fraction at least 50%
* Cardiac evaluation required if signs or symptoms of coronary artery disease or congestive heart failure

Other:

* HIV negative
* No active infection
* Patients excluded from this protocol are referred to protocol FHCRC-179.05

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1996-06; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Joachim Deeg, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Result] Anderson JE, Sale G, Appelbaum FR, Chauncey TR, Storb R. Allogeneic marrow transplantation for primary myelofibrosis and myelofibrosis secondary to polycythaemia vera or essential thrombocytosis. Br J Haematol. 1997 Sep;98(4):1010-6. doi: 10.1046/j.1365-2141.1997.3083125.x. PMID 9326205